CLINICAL TRIAL: NCT05604157
Title: Effect of Tourniquet on Local Tissue Concentrations of Cefazolin During Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: Ancef Dosage in Knee Arthroplasty : Tourniquet Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Adam Hart, Orthopaedic Surgeon, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-6782
Record Dates: First submitted 2022-06-22; First posted 2022-11-03 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Infections Joint Prosthetic
Keywords: Cefazolin; Tourniquet; Arthroplasty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tourniquet (Active Comparator): 25 participants with tourniquet application
  Interventions: Other: Use of Tourniquet
- No tourniquet (No Intervention): 25 participants without tourniquet application

INTERVENTIONS:
Other: Use of Tourniquet — Application of tourniquet or not in adults undergoing a primary total knee replacement.
  Arms: Tourniquet

SUMMARY:
Tourniquet inflation during total knee arthroplasty (TKA) is commonly used to reduce bleeding in the surgical field; thereby facilitating exposure and cementation. However, reducing circulation to the leg may also reduce antibiotic distribution to the peri-incisional tissues. Once inflated, further parenteral addition of antibiotics is not likely to achieve peak concentration. Some studies propose techniques of regional prophylaxis with a tourniquet to achieve higher cefazolin tissue concentrations. To our knowledge, the effect of tourniquet application on antibiotic tissue concentrations during total knee arthroplasty has not been explored. Furthermore, the effect of time from dose to incision, participants weight, and length of surgery on local tissue concentrations of Ancef are poorly understood. Considering that infections remain the leading source of early reoperation and revision surgery, insight and optimization of local tissue antibiotics is of paramount interest.

DETAILED DESCRIPTION:
In Canada, over 130 000 cases of primary joint arthroplasty are performed annually, and this number is increasing steadily with the aging population. Projections from the United States estimate that, by 2030, more than 3.5 million primary joint arthroplasties will be performed annually. Although rare, with reported rates of 0.5-2% within 2 years, periprosthetic joint infection (PJI) is a devastating complication with serious morbidity. Effective use of antibiotic prophylaxis remains an important measure to prevent progression of an intraoperative contamination of the surgical site to an overt clinical infection. It creates a hostile environment in blood and tissue inhibiting pathogens that could contaminate the wound throughout the procedure. In order to be effective, the concentration of antibiotic must exceed the minimum inhibitory concentration (MIC) of the organism between skin incision and wound closure. S. aureus and Coagulase-negative staphylocci (CoNS), including S.epidermidis, cause close to half of deep infections and reported MIC ranges from 0.5 to 8 ug/ml in bone. Achieving fourfold MIC in tissue is recommended for halting the pathogen Cefazolin, efficient against most common pathogens in orthopaedics, has a good tissue penetration, minimal toxicity, low cost, and therefore is the antibiotic of choice in arthroplasty procedures. Pharmacokinetics studies have showed that Cefazolin achieves peak bone concentrations 40 minutes after parenteral application and based on systemic dosage methods, guidelines recommend that the antibiotic should be infused within 60 minutes before surgical incision. Compared to conventional systemic dosing, modern techniques using liquid chromatography and mass spectrometry can adequately measure antibiotic concentration in tissue like fat and bone.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-85 who require a primary total knee replacement
* Any gender
* Osteoarthritis, rheumatoid arthritis, avascular necrosis

Exclusion Criteria:

* Severe allergy to antibiotic used in the study
* Severe renal dysfunction (eGFR < 30 ml/min)
* Methicillin-resistant Staphylococcus aureus (MRSA) colonization
* participants who require revision surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Local tissue concentrations of Cefazolin in serum, fat, synovium and bone | Two years for study completion
  The principle intervention in this study will be the application of a tourniquet or no tourniquet during the procedure and its effect on local tissue concentrations of Cefazolin

CONTACTS AND LOCATIONS:
Overall Officials: Adam Hart, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Dr, Adam Hart, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Bosco JA, Bookman J, Slover J, Edusei E, Levine B. Principles of Antibiotic Prophylaxis in Total Joint Arthroplasty: Current Concepts. J Am Acad Orthop Surg. 2015 Aug;23(8):e27-35. doi: 10.5435/JAAOS-D-15-00017. PMID 26209148
- [Background] Fletcher N, Sofianos D, Berkes MB, Obremskey WT. Prevention of perioperative infection. J Bone Joint Surg Am. 2007 Jul;89(7):1605-18. doi: 10.2106/JBJS.F.00901. No abstract available. PMID 17606802
- [Background] Bicanic G, Crnogaca K, Barbaric K, Delimar D. Cefazolin should be administered maximum 30 min before incision in total knee arthroplasty when tourniquet is used. Med Hypotheses. 2014 Jun;82(6):766-8. doi: 10.1016/j.mehy.2014.03.020. Epub 2014 Mar 25. PMID 24717822
- [Background] Burke JF. The effective period of preventive antibiotic action in experimental incisions and dermal lesions. Surgery. 1961 Jul;50:161-8. PMID 16722001
- [Background] Yamada K, Matsumoto K, Tokimura F, Okazaki H, Tanaka S. Are bone and serum cefazolin concentrations adequate for antimicrobial prophylaxis? Clin Orthop Relat Res. 2011 Dec;469(12):3486-94. doi: 10.1007/s11999-011-2111-8. Epub 2011 Oct 4. PMID 21968901
- [Background] Young SW, Zhang M, Freeman JT, Vince KG, Coleman B. Higher cefazolin concentrations with intraosseous regional prophylaxis in TKA. Clin Orthop Relat Res. 2013 Jan;471(1):244-9. doi: 10.1007/s11999-012-2469-2. PMID 22773397
- [Background] Bhalodi AA, Housman ST, Shepard A, Nugent J, Nicolau DP. Tissue pharmacokinetics of cefazolin in patients with lower limb infections. Antimicrob Agents Chemother. 2013 Nov;57(11):5679-83. doi: 10.1128/AAC.01348-13. Epub 2013 Sep 16. PMID 24041887
- [Background] Quintiliani R, Nightingale C. Principles of antibiotic usage. Clin Orthop Relat Res. 1984 Nov;(190):31-5. PMID 6488647
- [Background] Prokuski L, Clyburn TA, Evans RP, Moucha CS. Prophylactic antibiotics in orthopaedic surgery. Instr Course Lect. 2011;60:545-55. PMID 21553797
- [Background] Craig WA. Pharmacokinetic/pharmacodynamic parameters: rationale for antibacterial dosing of mice and men. Clin Infect Dis. 1998 Jan;26(1):1-10; quiz 11-2. doi: 10.1086/516284. PMID 9455502
- [Background] Steinberg JP, Braun BI, Hellinger WC, Kusek L, Bozikis MR, Bush AJ, Dellinger EP, Burke JP, Simmons B, Kritchevsky SB; Trial to Reduce Antimicrobial Prophylaxis Errors (TRAPE) Study Group. Timing of antimicrobial prophylaxis and the risk of surgical site infections: results from the Trial to Reduce Antimicrobial Prophylaxis Errors. Ann Surg. 2009 Jul;250(1):10-6. doi: 10.1097/SLA.0b013e3181ad5fca. PMID 19561486
- [Background] Zhang M, Moore GA, Chin PKL, Everts R, Begg EJ. Simultaneous Determination of Cefalexin, Cefazolin, Flucloxacillin, and Probenecid by Liquid Chromatography-Tandem Mass Spectrometry for Total and Unbound Concentrations in Human Plasma. Ther Drug Monit. 2018 Dec;40(6):682-692. doi: 10.1097/FTD.0000000000000555. PMID 30015652
- [Derived] Montreuil J, Tanzer M, Zhang YL, Rajda E, Avizonis D, Hart A. Tourniquet Use and Local Tissue Concentrations of Cefazolin During Total Knee Arthroplasty: A Randomized Clinical Trial. JAMA Netw Open. 2024 Aug 1;7(8):e2429702. doi: 10.1001/jamanetworkopen.2024.29702. PMID 39178000